CLINICAL TRIAL: NCT04297813
Title: Randomized Controlled Clinical Trial to Assess the Efficacy of a Combination of Autologous Mesenchymal Stem Cells and Biomaterial in Jaw Bone Regeneration Prior to Dental Implant Placement in Comparison to Standard Autologous Bone Grafting
Brief Title: Efficacy in Alveolar Bone Regeneration With Autologous MSCs and Biomaterial in Comparison to Autologous Bone Grafting
Acronym: Maxibone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Université de Nantes (Other); University of Ulm (Other); Universidad Complutense de Madrid (Other); University of Aarhus (Other); Universitat Internacional de Catalunya (Other); Assistance Publique - Hôpitaux de Paris (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001227-39; 2018-001227-39 (EudraCT Number)
Record Dates: First submitted 2020-02-25; First posted 2020-03-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2020-03

CONDITIONS: Alveolar Bone Atrophy
Keywords: Maxilla; mandible,; MSC; RCT; Bone regeneration; Multicenter
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Biocompatible Materials

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with advanced therapy medicinal product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): The gold standard; Bone block from the ramus of the nation will be transplanted to the alveolar ridge.
  Interventions: Procedure: Autologous bone graft
- Test (Experimental): Expanded, autologous mesenchymal stem cells in combination with biphasic calcium phosphate
  Interventions: Combination Product: Advanced medicinal Therapy (MSC combined with biomaterial)

INTERVENTIONS:
Combination Product: Advanced medicinal Therapy (MSC combined with biomaterial) — Augmentation of alveolar ridge with MSC and biomaterial
  Arms: Test
Procedure: Autologous bone graft — Augmentation of the alveolar ridge with bone graft
  Arms: Control

SUMMARY:
A randomized controlled clinical multi center trial to assess the efficacy of a combination of autologous mesenchymal stem cells and biomaterial in jaw bone regeneration prior to dental implant placement in comparison to standard autologous bone block grafting.

DETAILED DESCRIPTION:
A phase III multi center clinical trial, randomized and controlled.The study subject is lacking one or more sheet behind the canine in the upper or lower jaw, and the alveolar ridge is too narrow to place a dental implant. The test objects will have augmentation using autologous mesenchymal stromal cells and a biomaterial, biphasic Calcium Phosphate. The control is the traditional bone block from the ramus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non smoking patients in need of dental implants in the upper or lower jaw, with loss in vertical height and less that 4 mm in lateral width.

Exclusion Criteria:

* General contraindications for dental and/or surgical treatments
* Contraindications for both bone marrow harvesting and bone grafts
* History of any malignant diseases
* Concurrent or previous radiotherapy of head and neck region
* History of contagious diseases (HIV, HTLV and/or syphilis seropositivity, hepatitis B or C infection)
* Uncontrolled diabetes mellitis, e.g. patients with diabetes not regulated with medications or diet. This will be verified based on patient's history and concurrent HbA1c levels (HbA1c > 53 mmol/mol).
* Inflammatory and autoimmune disease of the oral cavity.
* Concurrent or previous immunosuppressant, bisphosphonate or high dose corticosteroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in bone width | 0-5 months
  Changes in linear measurements of bone width measured by CBCT.Principal assessment is linear change in bone width 2 mm below alveolar crest measured by means of CBCT images from baseline to 5 months after the regenerative surgery, immediately prior to implant placement

SECONDARY OUTCOMES:
Pain postoperatively in the two different treatments | 21 months
  Assessed by VAS scale, the scale goes from 0 to 100, 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
Radiological examination of bone volume | 21 months
  To evaluate the formation of the new bone by assessing if it is possible to insert an implant in the reconstructed area 5 months after the grafting procedure. This decision will be made based on radiological examination of bone volume by means of 3D CBCT images captured immediately prior to implant placement, 5-6 months after the regenerative surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Professor, Principal Investigator — Universidad Complutense de Madrid; Else Marie Pinholt, Professor, Principal Investigator — Syddansk Universitet SDU (University Hospital of Southern Denmark); Federico Hernandez-Alfaroo, Professor, Principal Investigator — Universitat Internacional de Catalunya; Alain Hoornaert, DDS, Principal Investigator — CHU Nantes, Centre de Soins Dentaires; Frederik Gaultier, PhD/DDS, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (6):
- Syddansk Universitet SDU (University Hospital of Southern Denmark), Odense, Denmark
- France (2):
  - Assistance Publique - Hôpitaux De Paris, Créteil
  - CHU Nantes, Centre de Soins Dentaires, Nantes
- University of Bergen, Institute of Clonical Dentistry, Bergen, Hordaland, Norway
- Spain (2):
  - Universidad Complutense De Madrid, Madrid, Calle Fernando de Castro Rodriguez,
  - Universitat Internacional De Catalunya, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement
URL: https://tissueengineering.no

REFERENCES:
- [Background] Gjerde C, Mustafa K, Hellem S, Rojewski M, Gjengedal H, Yassin MA, Feng X, Skaale S, Berge T, Rosen A, Shi XQ, Ahmed AB, Gjertsen BT, Schrezenmeier H, Layrolle P. Cell therapy induced regeneration of severely atrophied mandibular bone in a clinical trial. Stem Cell Res Ther. 2018 Aug 9;9(1):213. doi: 10.1186/s13287-018-0951-9. PMID 30092840
- [Background] Rojewski MT, Lotfi R, Gjerde C, Mustafa K, Veronesi E, Ahmed AB, Wiesneth M, Korper S, Sensebe L, Layrolle P, Hellem S, Schrezenmeier H. Translation of a standardized manufacturing protocol for mesenchymal stromal cells: A systematic comparison of validation and manufacturing data. Cytotherapy. 2019 Apr;21(4):468-482. doi: 10.1016/j.jcyt.2019.03.001. Epub 2019 Mar 27. PMID 30926359
- [Derived] Sanz M, Gjerde C, Gjertsen BT, Ortiz-Vigon A, Sanchez N, Hoornaert A, Caballe-Serrano J, Giralt-Hernando M, Gaultier F, Reinald N, Pinholt EM, Rojewski M, Rouard H, Chevallier N, Mohamed-Ahmed S, Shi X, Shi TJ, Schrezenmeier H, Layrolle P, Mustafa K. Bone Augmentation of Atrophic Alveolar Ridges Using a Synthetic Bone Substitute With Mesenchymal Stem Cells: A Randomized, Controlled Clinical Trial. Clin Oral Implants Res. 2025 Nov;36(11):1498-1514. doi: 10.1111/clr.70025. Epub 2025 Aug 22. PMID 40844304
- See also: Webpage for the clinical trial — https://tissueengineering.no